CLINICAL TRIAL: NCT06281470
Title: The First-in-Human, Single-Center, Randomized, Double-Blind, Placebo-Controlled，Single- and Multiple- Ascending Dose Study to Evaluate the Safety and Tolerability of WS016 in Healthy Chinese Volunteers
Brief Title: The Safety and Tolerability of WS016 in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Waterstone Pharmaceutical (Wuhan) Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WS016-Ⅰ-01
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Single Ascending Dose(SAD) Treatment 1 (Experimental): WS016 single dose（6g）
  Interventions: Drug: WS016 Single Dose(6g)
- SAD Treatment 2 (Experimental): WS016 single dose（12g）
  Interventions: Drug: WS016 Single Dose(12g)
- SAD Treatment 3 (Experimental): WS016 single dose（24g）
  Interventions: Drug: WS016 Single Dose(24g)
- SAD Treatment 4 (Experimental): WS016 single dose（36g）
  Interventions: Drug: WS016 Single Dose(36g)
- SAD Treatment 5 (Experimental): WS016 single dose（48g）
  Interventions: Drug: WS016 Single Dose(48g)
- SAD matching placebo (Placebo Comparator): SAD Matching placebo
  Interventions: Drug: SAD matching placebo
- Multiple Ascending Dose(MAD) Treatment 1 (Experimental): WS016 multiple dose(MAD Low Dose)
  Interventions: Drug: WS016 Multiple Dose(12g)
- MAD Treatment 2 (Experimental): WS016 multiple dose(MAD Medium Dose)
  Interventions: Drug: WS016 Multiple Dose(24g)
- MAD Treatment 3 (Experimental): WS016 multiple dose(MAD High Dose)
  Interventions: Drug: WS016 Multiple Dose(48g)
- MAD matching placebo (Placebo Comparator): MAD matching placebo
  Interventions: Drug: MAD matching placebo

INTERVENTIONS:
Drug: WS016 Single Dose(6g) — WS016 6g, to be administered orally as a single dose.
  Arms: Single Ascending Dose(SAD) Treatment 1
Drug: WS016 Single Dose(12g) — WS016 12g, to be administered orally as a single dose.
  Arms: SAD Treatment 2
Drug: WS016 Single Dose(24g) — WS016 24g, to be administered orally as a single dose.
  Arms: SAD Treatment 3
Drug: WS016 Single Dose(36g) — WS016 36g, to be administered orally as a single dose.
  Arms: SAD Treatment 4
Drug: WS016 Single Dose(48g) — WS016 48g, to be administered orally as a single dose.
  Arms: SAD Treatment 5
Drug: SAD matching placebo — Matching placebo, to be administered orally as a single dose.
  Arms: SAD matching placebo
Drug: WS016 Multiple Dose(12g) — WS016 12g, to be administered orally once daily for a consecutive period of 7 days.
  Arms: Multiple Ascending Dose(MAD) Treatment 1
Drug: WS016 Multiple Dose(24g) — WS016 24g, to be administered orally once daily for a consecutive period of 7 days.
  Arms: MAD Treatment 2
Drug: WS016 Multiple Dose(48g) — WS016 48g, to be administered orally once daily for a consecutive period of 7 days.
  Arms: MAD Treatment 3
Drug: MAD matching placebo — Matching placebo, to be administered orally once daily for a consecutive period of 7 days.
  Arms: MAD matching placebo

SUMMARY:
This clinic trial evaluates the safety and tolerability of single- and multiple- ascending doses of WS016 in healthy adult participants. There will be about 64 participants,48 active and 16 placebo.

ELIGIBILITY:
Inclusion Criteria:

1. The participants are fully informed of the purpose, methods and possible adverse reactions of the trial, and volunteer to serve as participants. And participants sign the informed consent form before any research procedures begin;
2. Participants are healthy male or female volunteers between the ages of 18 and 45 (including the cut-off values);
3. The weight of male participants is ≥50 kg, and the weight of female participants is ≥45 kg with a body mass index (BMI) of 19.0~26.0 kg/m^2 (including boundary values, BMI=weight (kg)/height^2 (m^2));
4. The participants understand and comply with the study procedures, can communicate well with the researchers, volunteer to participate in the trial, and sign the informed consent form.

Exclusion Criteria:

1. Participants with a specific allergy history (asthma, urticaria, eczema, etc.) or allergic constitution (e.g., known allergies to two or more substances), or known prior allergy to WS016 and related excipients;
2. Participants with chronic diseases or severe diseases in the liver, kidney, digestive system, endocrine system, cardiovascular system, nervous system, metabolic system, blood system, respiratory system, and autoimmune system, or current diseases in these systems as judged by investigators to be unsuitable for inclusion;
3. Participants who have undergone surgery within 3 months prior to screening, or plan to undergo surgery during the study period, as well as subjects who have undergone surgery that affects drug absorption, distribution, metabolism, and excretion;
4. Participants with dysphagia or gastrointestinal diseases/symptoms judged by investigators to affect drug absorption;
5. Participants who have received blood transfusions or used blood products ≥400 mL or 2 units within 3 months prior to screening, or have lost ≥400 mL of blood within 6 months, or have donated blood within 3 months;
6. Participants who have used any prescription drugs (including vaccines), over-the-counter drugs within 4 weeks prior to screening;
7. Pregnant or breastfeeding women, or participants with positive pregnancy test results before screening; male participants (or their partners) or female participants who have plans for pregnancy, sperm donation plans, or egg donation plans from the time they sign the informed consent form until 6 months after dosing; participants who are unwilling to use a medically recognized non-drug contraceptive method (e.g., intrauterine device or condom) during the study period;
8. Participants with abnormal findings in physical examination, vital signs examination, electrocardiogram, laboratory tests (including blood routine, urine routine, blood biochemistry, coagulation function), abdominal B-mode ultrasound examination, chest X-ray examination as judged by investigators to be clinically significant;
9. Participants with positive results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) quantitative test, human immunodeficiency virus (HIV) quantitative test, and syphilis antibody test;
10. Participants with a history of drug abuse within 12 months before screening, or urine drug screening positive results;
11. Participants with positive results in alcohol breath testing, or participants who consume alcohol regularly within 3 months before screening (defined as an average of more than 14 units of alcohol per week, and 1 unit is approximately equal to 200 mL of beer with a 5% alcohol content, or 25 mL of strong liquor with a 40% alcohol content, or 85 mL of wine with a 12% alcohol content), or participants who cannot abstain from alcohol during the study period;
12. Participants who are considered unsuitable for participation in this study by investigators.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Number of participants that experience Adverse Events (AEs) and Serious Adverse Events (SAEs) after single- and multiple- ascending dose | up to Day 17
  Incidence, severity and causality of AEs and SAEs

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Xiaoshan Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No